CLINICAL TRIAL: NCT03259711
Title: Cardiotoxicity of Selective Estrogen Receptor Modulators and Aromatase Inhibitors in the European Pharmacovigilance Database
Brief Title: Comparison of Cardiotoxicity Induced by Selective Estrogen REceptor Modulators and aNti-Aromatase
Acronym: SERENA
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-17-09
Record Dates: First submitted 2017-08-16; First posted 2017-08-24 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Affections
Keywords: Cardiotoxicity; selective estrogen receptor modulators; aromatase inhibitors; hormone replacement therapy; estrogen
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hormonal therapies L02 in the ATC classification — Hormonal therapies L02 in the ATC classification

SUMMARY:
Selective estrogen receptor modulators and aromatase inhibitors for the treatment of breast cancer seems to have an impact on the cardio-vascular system. This study investigates reports of cardiovascular toxicities for treatment including Anatomical Therapeutic Chemical (ATC) classification: L02 in the European pharmacovigilance database, Eudravigilance.

DETAILED DESCRIPTION:
Hormone replacement therapies and contraceptive pills are responsible of a wide range of cardio-vascular side effects, particularly thrombo-embolic disorders and ischemic heart disease. The difference of incidence and type of cardio-vascular events between men and women are strongly related to sex hormones. This study investigates the main characteristics of patients affected by cardiovascular side effects (of which ventricular arrhythmia's, QT prolongation and Torsade de Pointe) imputed to drugs classified as L02 according to ATC.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the Eudravigilance from 01/2002 to 08/2017
* Adverse event reported were including the MedDRA terms: SOC Cardiac Affections and the HLT Death and Sudden Death

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is selected in the Eurodravigilance database from 01/2002 to 08/2017 and included patients treated with hormonal therapies L02 in the ATC classification.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Analysis of disproportionality of reports for cardiotoxicity associated with selective estrogen receptor modulators as compared to aromatase inhibitors by performing a case- non-case study | Immediate evaluation

SECONDARY OUTCOMES:
Type of cardiotoxicity (ventricular arrhythmia's, QT prolongation and Torsade de Pointe) depending on the category and type of hormonal therapy (selective estrogen receptor modulators or aromatase inhibitors) | Immediate evaluation
Disproportionality analysis of the reporting of drug-induced ventricular arrhythmia's with selective estrogen receptor modulators as compared to aromatase inhibitors | Immediate evaluation
Disproportionality analysis of the reporting of drug- induced QT prolongation with selective estrogen receptor modulators as compared to aromatase inhibitors | Immediate evaluation
Disproportionality analysis of the reporting of drug-induced Torsade de Pointe with selective estrogen receptor modulators as compared to aromatase inhibitors | Immediate evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie Salem, MD, PhD, Principal Investigator — Centre Régional de Pharmaco-vigilance - Paris, Pitié-Salpétrière
Locations (1):
- Centre Régional de Pharmaco-vigilance - Paris, Pitié-Salpétrière, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Grouthier V, Lebrun-Vignes B, Glazer AM, Touraine P, Funck-Brentano C, Pariente A, Courtillot C, Bachelot A, Roden DM, Moslehi JJ, Salem JE. Increased long QT and torsade de pointes reporting on tamoxifen compared with aromatase inhibitors. Heart. 2018 Nov;104(22):1859-1863. doi: 10.1136/heartjnl-2017-312934. Epub 2018 May 2. PMID 29720397